CLINICAL TRIAL: NCT05856903
Title: Impact of Emicizumab on ACT (Activated Clotting Time) Using the i-STAT Alinity Analyzer: In Vitro Study in Severe Hemophiliacs A and Healthy Volunteers
Brief Title: Impact of Emicizumab on Activated Clotting Time Using the i-STAT Alinity Analyzer
Acronym: EMISTAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0124; 2023-A00897-38 (Other: ID RCB)
Record Dates: First submitted 2023-04-28; First posted 2023-05-12 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hemophilia A
Keywords: Activated Clotting Time; Hemophilia; Emicizumab
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe hemophiliac patients under emicizumab
  Interventions: Diagnostic Test: ACT
- Healthy volunteers
  Interventions: Diagnostic Test: ACT

INTERVENTIONS:
Diagnostic Test: ACT — ACT will be measured :
  * after in vitro spiking with unfractionated heparin of blood samples from severe hemophilia A patients already treated with emicizumab
  * after in vitro spiking with unfractionated heparin with or without emicizumab of blood samples from healthy volunteers

SUMMARY:
Emicizumab (Hemlibra®) is a subcutaneous hemostatic treatment approved in 2019 for the prophylaxis in severe hemophilia A. Emicizumab is a bispecific monoclonal antibody mimicking factor VIIIa that provides a constant level of coagulation similar to that observed in minor haemophilia A patients whose factor VIII level is 10-15%. Although the correction of plasma coagulation in vivo is only partial, emicizumab strongly shortens the in vitro coagulation times involving the intrinsic pathway such as aPTT(activated partial thromboplastin time).

The investigators will evaluate the effect of emicizumab on a coagulation test (Activating clotting time (ACT i-STAT Alinity)) used as a point of care device to monitor heparin therapies during cardiac surgeries (cardiopulmonary bypass) and cardiac catheterizations. Because ACT is activated through the intrinsic pathway, it may also be shortened by emicizumab. Prophylactic treatment with emicizumab would make it impossible to use ACT for heparin therapy in a hemophiliac patient benefiting from this treatment.

The aim of this in vitro study is to assess the effect of emicizumab on the in vitro heparin-induced ACT increase in severe hemophilia A patients treated with emicizumab and in healthy volunteers (measurement on the i- STAT Alinity) thanks to in vitro blood spiking experiments.

Some data have already been published with other ACT devices (Hemochron..) but never with the i-STAT Alinity device which uses a different technology and other reagents.

ELIGIBILITY:
Inclusion criteria:

* severe hemophiliacs under emicizumab ( > 4 weeks)

Exclusion Criteria:

* infusion of factor VIII < 5 days
* patients refusing to participate in the study
* protected persons
* anticoagulants

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: see above
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Modification of ACT by emicizumab | Day 0
  Modification of the in vitro heparin-induced ACT increase by emicizumab

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël MARLU, MD, Principal Investigator — Grenoble Alpes University Hospital
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mahlangu J, Oldenburg J, Paz-Priel I, Negrier C, Niggli M, Mancuso ME, Schmitt C, Jimenez-Yuste V, Kempton C, Dhalluin C, Callaghan MU, Bujan W, Shima M, Adamkewicz JI, Asikanius E, Levy GG, Kruse-Jarres R. Emicizumab Prophylaxis in Patients Who Have Hemophilia A without Inhibitors. N Engl J Med. 2018 Aug 30;379(9):811-822. doi: 10.1056/NEJMoa1803550. PMID 30157389
- [Background] Lenting PJ. Laboratory monitoring of hemophilia A treatments: new challenges. Blood Adv. 2020 May 12;4(9):2111-2118. doi: 10.1182/bloodadvances.2019000849. PMID 32396619
- [Background] Lowe A, Kitchen S, Jennings I, Kitchen DP, Woods TAL, Walker ID. Effects of Emicizumab on APTT, FVIII assays and FVIII Inhibitor assays using different reagents: Results of a UK NEQAS proficiency testing exercise. Haemophilia. 2020 Nov;26(6):1087-1091. doi: 10.1111/hae.14177. Epub 2020 Oct 23. PMID 33094895
- [Background] Wahba A, Milojevic M, Boer C, De Somer FMJJ, Gudbjartsson T, van den Goor J, Jones TJ, Lomivorotov V, Merkle F, Ranucci M, Kunst G, Puis L; EACTS/EACTA/EBCP Committee Reviewers. 2019 EACTS/EACTA/EBCP guidelines on cardiopulmonary bypass in adult cardiac surgery. Eur J Cardiothorac Surg. 2020 Feb 1;57(2):210-251. doi: 10.1093/ejcts/ezz267. No abstract available. PMID 31576396
- [Background] Capdevila L, Frere C, Desvages M, Harroche A, Bally C, Abbes A, d'Oiron R, Frenzel L, Borgel D, Lasne D. Emicizumab does not interfere with the activated clotting time. Haemophilia. 2022 Mar;28(2):362-366. doi: 10.1111/hae.14497. Epub 2022 Jan 21. PMID 35060654
- [Background] Isaacs J, Welsby IJ, Schroder JN, Onwuemene OA. Activated Coagulation Time and Hepcon Protamine Titration Device to Manage Unfractionated Heparin During Cardiopulmonary Bypass in a Hemophilia A Patient on Emicizumab. J Cardiothorac Vasc Anesth. 2021 Nov;35(11):3299-3302. doi: 10.1053/j.jvca.2020.08.058. Epub 2020 Aug 27. PMID 32928650